CLINICAL TRIAL: NCT06711068
Title: Cohort Study of Adjuvant Chemotherapy Combined With Targeted Therapy for Intermediate Risk HER2 Positive and Lymph Node Negative Early Breast Cancer
Brief Title: Adjuvant Therapy for Intermediate Risk HER2 Positive, Lymph Node Negative Early Breast Cancer With Chemotherapy Combined Target Therapy
Acronym: TaxDHER2
Status: Recruiting | Type: Observational
Sponsor: Shu Wang (Other)
Responsible Party: Sponsor-Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PKUPH2024Z165
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: HER2-positive Breast Cancer
Keywords: Taxane; target therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Taxanes combined with cyclophosphamide chemotherapy: Taxanes (paclitaxel, liposomal paclitaxel, docetaxel, albumin paclitaxel), cyclophosphamide chemotherapy, combined with targeted therapy with trastuzumab, for a total of 4 cycles, followed by targeted therapy maintenance for 1 year
- Taxanes chemotherapy: Taxanes (paclitaxel, liposomal paclitaxel, docetaxel, albumin paclitaxel) combined with trastuzumab and pertuzumab targeted therapy, for a total of 4 cycles, followed by targeted therapy maintenance for 1 year

SUMMARY:
Human epidermal growth factor receptor 2 (HER2) positive breast cancer is a molecular subtype with high malignancy and easy recurrence and metastasis. The emergence of HER2 targeted drugs has greatly improved the prognosis and survival of such patients. At present, for HER2 positive breast cancer patients with negative lymph nodes, chemotherapy drugs combined with trastuzumab is the current standard treatment scheme, and in most cases, chemotherapy uses a combination of two drugs, while the main beneficiaries of the trastuzumab and pertuzumab are concentrated in the group of patients with positive lymph nodes. Can targeted therapy be used to reduce the progression of chemotherapy and further achieve efficient and low toxicity strategies. It is planned to explore the efficacy and safety of T1-T2, HER2 positive early breast cancer patients with negative lymph nodes to achieve chemotherapy reduction based on risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* 1) Treatment in Peking University People's Hospital for radical resection of breast cancer and had hospitalization records;
* 2) Postoperative pathology confirmed invasive breast cancer, and the pathological stage was T1c, N0, HER2 positive, with other high-risk factors (G3, or hormone receptor negative); Or the pathological stage is T2, N0, and there are no high-risk factors (G3, or hormone receptor negative);
* 3)Signed an agreement to participate in the PKUPH Breast Disease Cohort study at Peking University People's Hospital.

Exclusion Criteria:

* 1) Lack of clinical pathological data (such as imaging data, pathological data);
* 2) Preoperative neoadjuvant therapy;
* 3) Patients with metastatic breast cancer or bilateral breast cancer;
* 4) Failed to undergo curative surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Invasive breast cancer, and the pathological stage was T1c, N0, HER2 positive, with other high-risk factors (G3, or hormone receptor negative); Or the pathological stage is T2, N0, and there are no high-risk factors (G3, or hormone receptor negative).
Sampling Method: Probability Sample
Enrollment: 8077 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 years
  The time from enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause.

SECONDARY OUTCOMES:
invasive disease free survival | 3 years
  The time from enrollment to the first occurrence of the following events defined as failure: local recurrence of ipsilateral invasive breast cancer, contralateral invasive breast cancer, distant recurrence or death from any cause.
distant disease free survival | 3 years
  The time from enrollment in the study to the occurrence of distant recurrence and metastasis
breast cancer specific survival | 3 years
  Time from enrollment to death due to breast cancer
overall survival | 3 years
  The time from enrollment in the study to death caused by any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China